CLINICAL TRIAL: NCT00758667
Title: Chemically Assisted Capsulectomy-A New Clinical Approach
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: preliminary analysis showed no difference
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, R. Bruce Shack, R. Bruce Shack, MD, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010518
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Implant Capsular Contracture
Keywords: capsular contracture; capsulectomy; mesna; Capsular contracture after breast implant placement
MeSH Terms: conditions — Implant Capsular Contracture | interventions — Mesna

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (No Intervention): Standard treatment
- Use of Mesna (Experimental): Standard surgical procedure with Mesna
  Interventions: Drug: Mesna

INTERVENTIONS:
Drug: Mesna — B. Mesna will be used to aid in the removal of the capsule when capsulectomy is performed
  Arms: Use of Mesna

SUMMARY:
The purpose of this study is to make available an agent,Mesna, which can assist the surgeon during the procedure of capsulectomy.

DETAILED DESCRIPTION:
Mesna is a FDA approved drug for the treatment of respiratory diseases and is used a protective agent against drugs in oncology patients. It has also been used in Gynecologic surgery and ENT. Mesna is a drug that breaks down adhesions between tissue layers.

ELIGIBILITY:
Inclusion Criteria:

* All females undergoing capsulectomy

Exclusion Criteria:

* All pregnant women and nursing mothers will be exclued

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shack, MD, Principal Investigator — Vanderbit Unviersity Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard: Standard procedure or capsulectomy for removal of capsule;
- Mesna: The use of Mesna of removal of capsule for capsular contracture.
  Mesna: A. Mesna will be used to aid in the removal of the capsule when capsulectomy is performed
Period: Overall Study
Arm/Group | Standard | Mesna
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with capsular contracture after breast implants that elected to have capsule removed and implant exchanged; followup for recurrence of capsulsar contracture
Groups:
- Standard: Standard procedure or capsulectomy for removal of capsule; no mesna
  Mesna: A. Mesna will be used to aid in the removal of the capsule when capsulectomy is performed
- Total: Total of all reporting groups
Arm/Group | Standard | Mesna | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Compare Number of Patients With Capsular Contracture in Mesna Group vs Standard of Care
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Standard | Mesna
Number analyzed (Participants) | 9 | 11
participants | 2 | 4

2. Secondary Outcome: Compare Number of Patients With Adverse Events in the Mesna Group vs the Standard of Care
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Standard | Mesna
Number analyzed (Participants) | 9 | 11
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | Standard | Mesna
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No